CLINICAL TRIAL: NCT02690324
Title: The Development of Skin Adhesive Patches for the Monitoring and Prediction of Mental Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-07-151
Record Dates: First submitted 2016-02-11; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2015-11

CONDITIONS: Major Depressive Disorder, Anxiety Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders

ARMS (3):
- Major depressive disorder (Experimental): DSM-5 major depressive disorder HAMD-17 > 16
  Interventions: Behavioral: cognitive stress (serial 7)
- panic disorder (Active Comparator): DSM-5 panic disorder PDSS>7
  Interventions: Behavioral: cognitive stress (serial 7)
- normal control (Active Comparator): age >20, healthy adults HAMD-17<17 PDSS<7
  Interventions: Behavioral: cognitive stress (serial 7)

INTERVENTIONS:
Behavioral: cognitive stress (serial 7)

SUMMARY:
development of skin adhesive patches for the monitoring and prediction of mental disorders

ELIGIBILITY:
Inclusion Criteria:

* the existence of a current Major depressive disorder or panic disorder during the screening and baseline visits, per the Mini-International Neuropsychiatric Interview (Sheehan et al., 1998) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* scored at least 16 on the HDRS-17 (Hamilton, 1960) for MDD and 7 on the Panic disorder severity scale for panic disorder patients at the baseline visits.

Exclusion Criteria:

* Patients who had psychotic disorder (e.g., schizophrenia or delusional disorder), bipolar affective disorder,active alcohol or drug use disorder, neurological illness including significant cognitive impairment or Parkinson's disease, mental retardation, significant medical conditions, epilepsy, histories of alcohol or drug dependence, personality disorders, or brain damages
* patients who were at serious risk for suicide of homicide

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Electrodermal activity(EDA) | baseline, 0.5, 1,2,3 months
  changes of skin conductane level(SCL) and skin conductance response(SCR)
Heart rate variability | baseline, 0.5, 1,2,3 months
  changes of SDNN, RMSSD and LF/HF ratio

SECONDARY OUTCOMES:
Brain-derived neurotrophic factor(BDNF) genotyping: Val66Met | baseline, 0.5, 1,2,3 months
Cytokines | baseline, 0.5, 1,2,3 months
  IL-1α, IL-1β, IL-2, IL-4, IL-6, IL-10, IL-12(p70), IFN-γ, TNF-α
Leptin | baseline, 0.5, 1,2,3 months
Adiponectin | baseline, 0.5, 1,2,3 months
Epinephrine | baseline, 0.5, 1,2,3 months
Norepinephrine | baseline, 0.5, 1,2,3 months
C reactive protein | baseline, 0.5, 1,2,3 months
BDNF | baseline, 0.5, 1,2,3 months
  serum, plasma, platelet BDNF
MINI plus | Baseline
  structured interview assessing for DSM-IV Axis I disorders with strong reliability and validity in relation to the Structured Clinical Interview for DSM-IV (SCID-IV)
MINI Suicidality Module | baseline, 0.5, 1,2,3 months
  assess current and past Axis I diagnoses
Hamilton Depression Rating Scale-17(HAMD-17) | baseline, 0.5, 1,2,3 months
  changes of HAMD-17 total socres
Hamilton Anxiety Rating Scale(HAMA) | baseline, 0.5, 1,2,3 months
  changes of HAMA total scores
Anxiety Sensitivity Index(ASI) | baseline, 0.5, 1,2,3 months
  ASI-3 to measure the three most supported AS domains: social (i.e., fear of exhibiting symptoms in public that may elicit embarrassment), cognitive (i.e., fear of losing cognitive control or experiencing concentration difficulties), and physical (i.e., fear that physical sensations are a sign of an immediate physical problem).
APPQ(Albany Panic and Phobia Questionnaire) | baseline, 0.5, 1,2,3 months
  The APPQ (Rapee et al., 1995) is a 27-item instrument that is designed to measure interoceptive, agoraphobic, and social situational fear. Subjects respond to each item on a 9-point Likert scale from 0 to 8, according to how much fear they think they would experience in a given situation so that total scores range from 0 to 216.
PSWQ(Penn state worry questionnaire) | baseline, 0.5, 1,2,3 months
  16-item questionnaire that aims to measure the trait of worry, using Likert rating from 1 (not at all typical of me) to 5 (very typical of me)
SRI(Stress response Inventory) | baseline, 0.5, 1,2,3 months
  emotional, somatic, cognitive, and behavioral stress responses.
Perceived Stress Scale(PSS) | baseline, 0.5, 1,2,3 months
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful.
Barratt Impulsivity Scale | baseline, 0.5, 1,2,3 months
  The Barratt Impulsiveness Scale (BIS) is a widely used measure of impulsiveness. It includes 30 items that are scored to yield six first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and three second-order factors (attentional, motor, and non-planning impulsiveness).The BIS-11 is a 30-item self-report questionnaire, that is scored to yield a total score, three second-order factors, and six first-order factors.
Panic disorder severity scale(PDSS) | baseline, 0.5, 1,2,3 months
  The items assess panic frequency, distress during panic, panic-focused anticipatory anxiety, phobic avoidance of situations, phobic avoidance of physical sensations, impairment in work functioning, and impairment in social functioning. The overall assessment is made by a total score, which is calculated by summing the scores for all seven items. The total scores range from 0 to 28.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Irwon-dong, Gangnam-gu, South Korea